CLINICAL TRIAL: NCT00428272
Title: A Phase I Trial of Monoclonal Antibody HGS-ETR2 (Lexatumumab) With or Without Interferon Gamma in Patients With Refractory Pediatric Solid Tumors
Brief Title: HGS-ETR2 to Treat Children With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070040; 07-C-0040; NCT01445093 (obsolete NCT alias)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-10-09

CONDITIONS: Ewing's Sarcoma; Osteosarcoma; Neuroblastoma; Rhabdomyosarcoma
Keywords: Monoclonal Antibody Lexatumumab; Interferon Gamma; Solid Tumor; Phase I; Malignant Tumor; Metastatic Tumor; Pediatric Solid Tumor; Ewing Sarcoma; Osteosarcoma; Neuroblastoma; Rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma; Neuroblastoma; Rhabdomyosarcoma; Neoplasms; Neoplasm Metastasis | interventions — lexatumumab; Interferon-gamma

ARMS (3):
- 1 (Experimental): Lexatumumab alone dose escalation
  Interventions: Drug: Lexatumumab alone
- 2 (Experimental): Lexatumumab with interferon - dose escalation
  Interventions: Drug: Lexatumumab in combination; Drug: Interferon gamma 1b in combination
- 3 (Other): Lexatumumab 10mg/kg with interferon expansion at
  Interventions: Drug: Lexatumumab in combination; Drug: Gamma 1b potential expansion

INTERVENTIONS:
Drug: Lexatumumab alone — Dose escalation : 3mg/kg, 5mg/kg, 8mg/kg, 10mg/kg
  Arms: 1
Drug: Lexatumumab in combination — Dose escalation : 1mg/kg, 3mg/kg, 5mg/kg, 8mg/kg, 10mg/kg
  Arms: 2; 3
Drug: Interferon gamma 1b in combination — Dosing at the following for each lexatumumab dose level: .75mcg/m2/dose and 25mcg/m2/dose
  Arms: 2
Drug: Gamma 1b potential expansion — Potential expansion (at 10mg/kg lexatumumab): 1.5mcg/m2/dose and 50mcg/m2/dose
  Arms: 3

SUMMARY:
Background

* HGS-ETR2 is a monoclonal antibody, produced in the laboratory from human genes.
* HGS-ETR2 targets a protein called the TRAIL receptor that is located on the surface of some tumor cells. When the TRAIL receptor is activated, it can cause the tumor cell to self-destruct.

Objectives:

* To determine the highest dose of HGS-ETR2 that can be given safely in children and young adults with cancer.
* To study the pharmacology (how the body handles the drug) of HGS-ETR2 by measuring the amount of drug in the bloodstream over time before and after a dose is given to the patient.
* To determine if HGS-ETR2 can stop or slow tumor growth.
* To determine whether proteins in tumor tissue before treatment can predict whether the tumor will respond to HGS-ETR2 therapy.

Eligibility:

-Patients 1 to 21 years of age with solid cancers that do not respond to standard therapy.

Design:

* HGS-ETR2 is given through a vein (intravenously, IV) once every 14 days. Each treatment cycle is 28 days long and consists of two doses of HGS-ETR2.
* The dose of HGS-ETR2 is increased in successive small groups of patients until the maximum tolerated dose (highest dose with acceptable side effects) is determined.
* During the treatment period, patients have a physical examination at least once a week, and routine blood tests at least twice a week. These tests are done less frequently in later treatment cycles.
* Additional blood samples are drawn for immunology and pharmacology studies.
* Tests to monitor the size of the tumor (X-rays, CT scans, MRI, PET scans) are done periodically throughout the treatment period.
* Patients may continue to receive HGS-ETR2 until unacceptable side effects develop or the tumor grows.

DETAILED DESCRIPTION:
Background:

Pediatric solid tumors represent approximately one fourth of cancer diagnoses in children. Despite intensive regimens, patients with metastatic or recurrent tumors have unsatisfactory survival rates. Therefore new therapies are needed to improve outcomes.

Members of the TNF ligand superfamily induce death in tumor cells through direct ligation of death receptors and apoptosis induction.

TRAIL (TNF-related apoptosis inducing ligand) has specific anti-tumor activity against a wide range of tumor cells without inducing death in normal cells. TRAIL-induced apoptosis has been demonstrated in a wide variety of pediatric solid tumors, including Ewing's sarcoma, osteosarcoma, neuroblastoma, and rhabdomyosarcoma.

HGS-ETR2 (Human Genome Sciences; human monoclonal antibody) is a fully human monoclonal antibody that agonistically binds TRAIL receptor 2 and, like TRAIL itself, induces apoptosis in a variety of malignant cell types with little effect on normal cells.

Limited caspase 8 expression is a primary factor in limiting to TRAIL mediated cell death in some tumors; interferon gamma has been shown to be effective in increasing caspase-8 expression in tumors and in restoring sensitivity of tumors to TRAIL mediated cell death.

Objectives:

To determine the tolerance of the adult maximum tolerated dose and dose limiting toxicities of lexatumumab in patients with refractory pediatric solid tumors.

To determine the MTD of lexatumumab in the presence of fixed dosing of interferon gamma 1b at 25 mcg/m(2) SC three times/week, which is less than the FDA approved dose.

To assess the pharmacokinetics of lexatumumab or lexatumumab in combination with interferon gamma 1b in patients with pediatric malignant tumors refractory to standard therapy.

Eligibility:

Patients must be 1-30 years of age with solid malignant tumors refractory to standard therapy.

Design:

A Phase I dose escalation study with 4 planned dose levels of lexatumumab starting at 30% of the adult MTD and escalating up to 100% of the adult MTD, followed by a second dose escalation using five lexatumumab dose levels in patients concomitantly receiving interferon gamma 1b.

Three (expanded to six if DLT occurs) patients will be enrolled at each dose level of lexatumumab until the adult MTD is reached and 6 patients will be enrolled at the adult MTD dose. The MTD cohort of lexatumumab alone and combined regimen will be expanded to include 12 patients, which should include a minimum of 6 patients less than or equal to 12 years of age. Once 6 patients greater than 12 years of age have completed lexatumumab alone, new patients greater than 12 years of age will be enrolled in the combined regimen. Similarly, once 6 patients complete lexatumumab alone who are less than or equal to 12 years of age, new patients less than or equal to 12 years of age will be enrolled in the combined regimen. A final dose escalation of interferon gamma 1b will be performed with the maximum dose level of lexatumumab, to a dose level wherein archival tissue demonstrated upregulation of caspase 8.

ELIGIBILITY:
* INCLUSION CRITERIA:

AGE: Patients must be greater than or equal to 1 years and less than or equal to 30 years of age in order to encompass a broad range of ages in children as well as to capture the young adult population which is highly represented in many of these types of sarcomas being studied.

DIAGNOSIS: Histologically confirmed solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing s sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilm s tumor, Hodgkin's or non-Hodgkin's lymphoma. Patients with primary or untreated metastatic CNS tumors or primary or metastatic hepatic tumors will not be treated on this study.

MEASURABLE/EVALUABLE DISEASE: Patients must have measurable or evaluable tumors.

PRIOR THERAPY:

The patient s cancer must have relapsed following or failed to respond to standard therapy, and the patient s current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.

Patients must have completed their last dose of irradiation, chemotherapy, monoclonal antibody, or investigational therapy at least 4 weeks prior to enrollment or their last dose of nitrosurea (CCNU, BCNU) 6 weeks prior to enrollment. For patients who have undergone autologous stem cell transplantation, at least 3 months must have elapsed since transplant.

Patients must have recovered from the toxic effects of all prior therapy prior to enrollment.

Patients must have been off colony stimulating factors (e.g. G-CSF, GM-CSF, Epo) for at least 72 hours prior to enrollment.

Patients must have completed any biological therapy (including investigational therapies) at least 7 days prior to study entry.

PERFORMANCE STATUS: Patients greater than 10 years old must have a Karnofsky Score of greater than or equal to 50 and children less than or equal to 10 years old must have a Lansky score of greater than 50. Patients who are unable to walk because of paralysis or weakness, but who are up in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.

HEMATOLOGIC FUNCTION: Patients must have adequate bone marrow function, defined as a peripheral absolute granulocyte count of greater than or equal to 1000/microliter, hemoglobin greater than or equal to 8 gm/dl, and a transfusion independent platelet count greater than or equal to 75,000/microliter.

Cardiac Function: Patients must have an ejection fraction of greater than 40% via MUGA or Echo or a shortening fraction greater than 27% by Echo and must not have had a history of congestive heart failure.

HEPATIC FUNCTION: Aspartate transaminase (AST) and alanine transaminase (ALT), less than or equal to 2.5-fold the upper limit of normal (ULN). Direct bilirubin within normal limits.

RENAL FUNCTION: Patients must have normal age-adjusted serum creatinine (see Table below) OR a creatinine clearance greater than or equal to 60 mL/min/1.73 m(2).

Age Less than or equal to 5 with a max serum creatinine (mg/dl) of 0.8

Age less than 5 less than or equal to 10 with a max serum creatinine (mg/dl) of 1.0

Age less than 10 less than or equal to 15 with a max serum creatinine (mg/dl) of 1.2

Less than 15 with a max serum creatinine (mg/dl) of 1.5

INFORMED CONSENT: All patients or their legal guardians (if the patients is less than18 years old) must sign a document of informed consent (Pediatric Oncology Branch, NCI screening protocol for NIH patients) prior to performing studies to determine patient eligibility. After confirmation of eligibility, all patients or their legal guardians must voluntarily sign the IRB approved protocol specific informed

this study and their willingness to receive the therapy and to undergo the research studies involved including pharmacokinetic studies. The consent must be signed before any protocol related studies are performed (This does not include routine laboratory tests or imaging studies required to establish eligibility). When appropriate, pediatric patients will be included in all discussions in order to obtain verbal assent. Assent will be obtained according to local IRB requirements.

DURABLE POWER OF ATTORNEY (DPA): Patients who are greater than or equal to 18 years of age will be offered the opportunity to assign a DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

BIRTH CONTROL: Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study and for 60 days following the last dose.

EXCLUSION CRITERIA:

Clinically significant unrelated systemic illness, such as serious infections or organ dysfunction, which in the judgment of the Principal or Associate Investigators would compromise the patient s ability to tolerate the agents in this trial or are likely to interfere with the study procedures or results.

Patients with a history of allogeneic bone marrow transplantation. Patients who have received autologous stem cell transplantation are eligible greater than 3 months after completion of therapy if they meet other eligibility requirements.

Patients with hepatic tumors or metastases are excluded due to the potential for hepatotoxicity with agents that target the TRAIL-R pathway. Patients with primary CNS tumors will be excluded due to unknown penetration into the CNS.

Untreated CNS metastases will render the patient ineligible however patients with a previous history of CNS metastases are eligible if: the metastases have been treated with surgery and/or radiotherapy, are clinically stable as evidenced by no requirements for corticosteroids, the patient has no evolving neurologic deficits and no change in residual brain abnormalities without specific therapy over 6 weeks.

Pregnant or breastfeeding females are excluded because the risks of lexatumumab to the developing fetus or nursing child are unknown.

Patients currently receiving other investigational agents.

History of any infection requiring hospitalization or parenteral antibiotics within 2 weeks of study entry.

Co-existing medical illness that would place the subject at undue risk.

On immunosupressant therapy (with the exception of prednisone up to 10 mg/day, or dexamethasone up to 4 mg/day), or with known human immunodeficiency virus (HIV) infection or hepatitis B or C. Subjects with immune deficiency are excluded due to their increased risk of life threatening toxicity when treated with anticancer agents.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12-04; Primary Completion 2011-04-28 (Actual); Study Completion 2015-10-09 (Actual)

PRIMARY OUTCOMES:
Asult MTD and DLTs of lexatumumab | 6 months
MTD of lexatumumab w/interferon gamma 1b | 6 months
Pharmacokinetics | 2 years

SECONDARY OUTCOMES:
Tumor response rate | 2 years
Correlation of immunohistochemical expression of pro-apoptotic proteins with response to therapy | 2 years
Determine if anti-HGS-ETR2 antibodies are produced | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Mackall, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wiley SR, Schooley K, Smolak PJ, Din WS, Huang CP, Nicholl JK, Sutherland GR, Smith TD, Rauch C, Smith CA, et al. Identification and characterization of a new member of the TNF family that induces apoptosis. Immunity. 1995 Dec;3(6):673-82. doi: 10.1016/1074-7613(95)90057-8. PMID 8777713
- [Background] Georgakis GV, Li Y, Humphreys R, Andreeff M, O'Brien S, Younes M, Carbone A, Albert V, Younes A. Activity of selective fully human agonistic antibodies to the TRAIL death receptors TRAIL-R1 and TRAIL-R2 in primary and cultured lymphoma cells: induction of apoptosis and enhancement of doxorubicin- and bortezomib-induced cell death. Br J Haematol. 2005 Aug;130(4):501-10. doi: 10.1111/j.1365-2141.2005.05656.x. PMID 16098063
- [Background] Younes M, Georgakis GV, Rahmani M, Beer D, Younes A. Functional expression of TRAIL receptors TRAIL-R1 and TRAIL-R2 in esophageal adenocarcinoma. Eur J Cancer. 2006 Mar;42(4):542-7. doi: 10.1016/j.ejca.2005.11.013. Epub 2006 Jan 19. PMID 16426839
- [Derived] Merchant MS, Geller JI, Baird K, Chou AJ, Galli S, Charles A, Amaoko M, Rhee EH, Price A, Wexler LH, Meyers PA, Widemann BC, Tsokos M, Mackall CL. Phase I trial and pharmacokinetic study of lexatumumab in pediatric patients with solid tumors. J Clin Oncol. 2012 Nov 20;30(33):4141-7. doi: 10.1200/JCO.2012.44.1055. Epub 2012 Oct 15. PMID 23071222